CLINICAL TRIAL: NCT00749658
Title: Human Laboratory Study of Varenicline and Bupropion for Nicotine Dependence
Acronym: ChanBan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCRC 10047; K01DA019446 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Nicotine Dependence; Nicotine Withdrawal
Keywords: Tobacco; Nicotine; Smoking; Varenicline; Bupropion; Human laboratory study; Stress tolerance; Startle response; Cognitive assessment; Progressive ratio; Motivation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Bupropion; Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion + Placebo Varenicline (Active Comparator): Bupropion + Placebo Varenicline \Varenicline + Placebo Bupropion; Varenicline + Placebo Bupropion \Bupropion + Placebo Varenicline
  Interventions: Drug: Bupropion; Drug: Varenicline
- upropion + Varenicline (Active Comparator): Bupropion + Varenicline \Varenicline + Placebo Bupropion; Varenicline + Placebo Bupropion \Bupropion + Varenicline
  Interventions: Drug: Bupropion; Drug: Varenicline

INTERVENTIONS:
Drug: Bupropion — Form: tablet, Dosage, Frequency, Duration: Days 1-3, 150 mg, q.d., Days 4-11, 150 mg, b.i.d.
  Other Names: Zyban; Wellbutrin
Drug: Varenicline — Form: tablet, Dosage, Frequency, Duration: Days 1-3, .5 mg, q.d., Days 4-7, .5 mg, b.i.d., Days 8-11, 1 mg, b.i.d.
  Other Names: Chantix

SUMMARY:
The objective of this proposal is to elucidate effects of bupropion SR + varenicline on smoking-cessation related processes in early abstinence using a human laboratory model. A within-subjects design will be used to assess the additive effects of bupropion and varenicline in 48 treatment seeking smokers [bupropion SR (300 mg/day)+placebo, varenicline (2 mg/day+placebo, and bupropion SR (300 mg/day)+varenicline (2 mg/day)]. Outcomes include withdrawal and craving, cognition, stress tolerance, anxiety, the reinforcing effects of smoking, and smoking topography.

Hypotheses: We hypothesize that greatest treatment effects will be observed in the bupropion SR+varenicline group followed by varenicline+placebo and bupropion SR+placebo groups.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and up.
2. Smoked at least 10 cigarettes/day for at least 1 year.
3. English speaking and reading.
4. Females who are of childbearing potential must practice effective contraception and meet the following criteria:

   1. Are instructed to avoid pregnancy through 30 days after the last dose of study medication.
   2. Have a negative urine pregnancy test at baseline.
   3. Agree to use of the birth control methods listed: an oral contraceptive agent, an intrauterine device (IUD), an implantable contraceptive (e.g., Norplant), or an injectable contraceptive (e.g., Depo-Provera) for at least one month prior to entering the study and will continue its use through at least 30 days after the last dose of the study medication. A barrier method of contraception (e.g., condom or diaphragm with spermicide) while participating in the study and 30 days after the last dose of study medication.
5. Willingness to not use illicit drugs during study period including marijuana.

Exclusion Criteria:

1. Any unstable medical condition.
2. Unstable angina, myocardial infarction, or coronary angioplasty within the past 3 months or an untreated cardiac dysrhythmia.
3. Personal history of seizures.
4. Closed head trauma with any loss of consciousness or amnesia in the last 5 years.
5. A history of closed head trauma with > 30 minutes of loss of consciousness or amnesia or resulting in skull fracture or subdural hematoma/brain contusion.
6. A history of psychosis, bipolar disorder, bulimia or anorexia nervosa.
7. Current depression as assessed by Center for Epidemiologic Studies Depression Scale (CES-D).
8. Medications that might affect the outcome measures of nicotine reward, cognition, anxiety, and stress will also be a basis for exclusion. These medications include psychotropic drugs (i.e., anti-psychotic, anti-depressant, anti-anxiety, or stimulant), anti- hypertensive agents (e.g., beta-blockers), and other drugs that can influence the outcome domains.
9. Active substance abuse other than nicotine.
10. Used an investigational drug within the last 30 days.
11. Are currently using a behavioral or pharmacologic tobacco treatment.
12. Use of bupropion or varenicline in the previous 30 days.
13. Current (past 14 days) use of antipsychotic or antidepressant medications.
14. An allergy to bupropion or varenicline.
15. Untreated hypertension or baseline systolic blood pressure > 180 or diastolic > 100.
16. Impaired kidney function (creatinine clearance < 30).
17. Having plans to leave the immediate geographical area within 2 months.
18. Unwillingness or inability to give written informed consent.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Mooney, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Tobacco Use Research Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ingersoll KS, Cohen J. Combination treatment for nicotine dependence: state of the science. Subst Use Misuse. 2005;40(13-14):1923-43, 2043-8. doi: 10.1080/10826080500294817. PMID 16282086
- [Background] Sweeney CT, Fant RV, Fagerstrom KO, McGovern JF, Henningfield JE. Combination nicotine replacement therapy for smoking cessation: rationale, efficacy and tolerability. CNS Drugs. 2001;15(6):453-67. doi: 10.2165/00023210-200115060-00004. PMID 11524024
- [Background] Biberman R, Neumann R, Katzir I, Gerber Y. A randomized controlled trial of oral selegiline plus nicotine skin patch compared with placebo plus nicotine skin patch for smoking cessation. Addiction. 2003 Oct;98(10):1403-7. doi: 10.1046/j.1360-0443.2003.00524.x. PMID 14519177
- [Background] Bohadana A, Nilsson F, Rasmussen T, Martinet Y. Nicotine inhaler and nicotine patch as a combination therapy for smoking cessation: a randomized, double-blind, placebo-controlled trial. Arch Intern Med. 2000 Nov 13;160(20):3128-34. doi: 10.1001/archinte.160.20.3128. PMID 11074742
- [Background] Cinciripini PM, Tsoh JY, Wetter DW, Lam C, de Moor C, Cinciripini L, Baile W, Anderson C, Minna JD. Combined effects of venlafaxine, nicotine replacement, and brief counseling on smoking cessation. Exp Clin Psychopharmacol. 2005 Nov;13(4):282-92. doi: 10.1037/1064-1297.13.4.282. PMID 16366758
- [Background] Croghan GA, Sloan JA, Croghan IT, Novotny P, Hurt RD, DeKrey WL, Mailliard JA, Ebbert LP, Swan DK, Walsh DJ, Wiesenfeld M, Levitt R, Stella P, Johnson PA, Tschetter LK, Loprinzi C. Comparison of nicotine patch alone versus nicotine nasal spray alone versus a combination for treating smokers: a minimal intervention, randomized multicenter trial in a nonspecialized setting. Nicotine Tob Res. 2003 Apr;5(2):181-7. doi: 10.1080/1462220031000073252. PMID 12745490
- [Background] Croghan IT, Hurt RD, Dakhil SR, Croghan GA, Sloan JA, Novotny PJ, Rowland KM, Bernath A, Loots ML, Le-Lindqwister NA, Tschetter LK, Garneau SC, Flynn KA, Ebbert LP, Wender DB, Loprinzi CL. Randomized comparison of a nicotine inhaler and bupropion for smoking cessation and relapse prevention. Mayo Clin Proc. 2007 Feb;82(2):186-95. doi: 10.4065/82.2.186. PMID 17290726
- [Background] Evins AE, Cather C, Culhane MA, Birnbaum A, Horowitz J, Hsieh E, Freudenreich O, Henderson DC, Schoenfeld DA, Rigotti NA, Goff DC. A 12-week double-blind, placebo-controlled study of bupropion sr added to high-dose dual nicotine replacement therapy for smoking cessation or reduction in schizophrenia. J Clin Psychopharmacol. 2007 Aug;27(4):380-6. doi: 10.1097/01.jcp.0b013e3180ca86fa. PMID 17632223
- [Background] Fagerstrom KO, Tonnesen P. Nicotine chewing gum and nicotine patch. Wien Med Wochenschr. 1995;145(4):77-82. PMID 7778323
- [Background] Hall SM, Humfleet GL, Reus VI, Munoz RF, Cullen J. Extended nortriptyline and psychological treatment for cigarette smoking. Am J Psychiatry. 2004 Nov;161(11):2100-7. doi: 10.1176/appi.ajp.161.11.2100. PMID 15514412
- [Background] Jorenby DE, Leischow SJ, Nides MA, Rennard SI, Johnston JA, Hughes AR, Smith SS, Muramoto ML, Daughton DM, Doan K, Fiore MC, Baker TB. A controlled trial of sustained-release bupropion, a nicotine patch, or both for smoking cessation. N Engl J Med. 1999 Mar 4;340(9):685-91. doi: 10.1056/NEJM199903043400903. PMID 10053177
- [Background] Killen JD, Fortmann SP, Schatzberg AF, Hayward C, Sussman L, Rothman M, Strausberg L, Varady A. Nicotine patch and paroxetine for smoking cessation. J Consult Clin Psychol. 2000 Oct;68(5):883-9. PMID 11068974
- [Background] Killen JD, Robinson TN, Ammerman S, Hayward C, Rogers J, Stone C, Samuels D, Levin SK, Green S, Schatzberg AF. Randomized clinical trial of the efficacy of bupropion combined with nicotine patch in the treatment of adolescent smokers. J Consult Clin Psychol. 2004 Aug;72(4):729-35. doi: 10.1037/0022-006X.72.4.729. PMID 15301658
- [Background] Kornitzer M, Boutsen M, Dramaix M, Thijs J, Gustavsson G. Combined use of nicotine patch and gum in smoking cessation: a placebo-controlled clinical trial. Prev Med. 1995 Jan;24(1):41-7. doi: 10.1006/pmed.1995.1006. PMID 7740014
- [Background] Krishnan-Sarin S, Meandzija B, O'Malley S. Naltrexone and nicotine patch smoking cessation: a preliminary study. Nicotine Tob Res. 2003 Dec;5(6):851-7. doi: 10.1080/14622200310001614601. PMID 14750508
- [Background] O'Malley SS, Cooney JL, Krishnan-Sarin S, Dubin JA, McKee SA, Cooney NL, Blakeslee A, Meandzija B, Romano-Dahlgard D, Wu R, Makuch R, Jatlow P. A controlled trial of naltrexone augmentation of nicotine replacement therapy for smoking cessation. Arch Intern Med. 2006 Mar 27;166(6):667-74. doi: 10.1001/archinte.166.6.667. PMID 16567607
- [Background] Piper ME, Federman EB, McCarthy DE, Bolt DM, Smith SS, Fiore MC, Baker TB. Efficacy of bupropion alone and in combination with nicotine gum. Nicotine Tob Res. 2007 Sep;9(9):947-54. doi: 10.1080/14622200701540820. PMID 17763111
- [Background] Rose JE, Behm FM, Westman EC. Nicotine-mecamylamine treatment for smoking cessation: the role of pre-cessation therapy. Exp Clin Psychopharmacol. 1998 Aug;6(3):331-43. doi: 10.1037//1064-1297.6.3.331. PMID 9725117
- [Background] Williams J, Ziedonis DM. Naltrexone-bupropion combination therapy for protracted abstinence dysphoria. Am J Addict. 2003 May-Jun;12(3):270-2. No abstract available. PMID 12851023
- [Background] Rose JE, Levin ED. Concurrent agonist-antagonist administration for the analysis and treatment of drug dependence. Pharmacol Biochem Behav. 1992 Jan;41(1):219-26. doi: 10.1016/0091-3057(92)90086-u. PMID 1539072
- [Background] Ascher JA, Cole JO, Colin JN, Feighner JP, Ferris RM, Fibiger HC, Golden RN, Martin P, Potter WZ, Richelson E, et al. Bupropion: a review of its mechanism of antidepressant activity. J Clin Psychiatry. 1995 Sep;56(9):395-401. PMID 7665537
- [Background] Coe JW, Brooks PR, Vetelino MG, Wirtz MC, Arnold EP, Huang J, Sands SB, Davis TI, Lebel LA, Fox CB, Shrikhande A, Heym JH, Schaeffer E, Rollema H, Lu Y, Mansbach RS, Chambers LK, Rovetti CC, Schulz DW, Tingley FD 3rd, O'Neill BT. Varenicline: an alpha4beta2 nicotinic receptor partial agonist for smoking cessation. J Med Chem. 2005 May 19;48(10):3474-7. doi: 10.1021/jm050069n. PMID 15887955
- [Background] Mooney ME, Sofuoglu M. Bupropion for the treatment of nicotine withdrawal and craving. Expert Rev Neurother. 2006 Jul;6(7):965-81. doi: 10.1586/14737175.6.7.965. PMID 16831112
- [Background] Warner C, Shoaib M. How does bupropion work as a smoking cessation aid? Addict Biol. 2005 Sep;10(3):219-31. doi: 10.1080/13556210500222670. PMID 16109583
- [Background] Johnston AJ, Ascher J, Leadbetter R, Schmith VD, Patel DK, Durcan M, Bentley B. Pharmacokinetic optimisation of sustained-release bupropion for smoking cessation. Drugs. 2002;62 Suppl 2:11-24. doi: 10.2165/00003495-200262002-00002. PMID 12109932
- [Background] Bondarev ML, Bondareva TS, Young R, Glennon RA. Behavioral and biochemical investigations of bupropion metabolites. Eur J Pharmacol. 2003 Aug 1;474(1):85-93. doi: 10.1016/s0014-2999(03)02010-7. PMID 12909199
- [Background] Hughes JR, Keely JP, Niaura RS, Ossip-Klein DJ, Richmond RL, Swan GE. Measures of abstinence in clinical trials: issues and recommendations. Nicotine Tob Res. 2003 Feb;5(1):13-25. PMID 12745503
- [Background] SRNT Subcommittee on Biochemical Verification. Biochemical verification of tobacco use and cessation. Nicotine Tob Res. 2002 May;4(2):149-59. doi: 10.1080/14622200210123581. No abstract available. PMID 12028847
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Shiffman S, Johnston JA, Khayrallah M, Elash CA, Gwaltney CJ, Paty JA, Gnys M, Evoniuk G, DeVeaugh-Geiss J. The effect of bupropion on nicotine craving and withdrawal. Psychopharmacology (Berl). 2000 Jan;148(1):33-40. doi: 10.1007/s002130050022. PMID 10663415
- [Background] Kotlyar M, Brauer LH, al'absi M, Adson DE, Robiner W, Thuras P, Harris J, Finocchi ME, Bronars CA, Candell S, Hatsukami DK. Effect of bupropion on physiological measures of stress in smokers during nicotine withdrawal. Pharmacol Biochem Behav. 2006 Mar;83(3):370-9. doi: 10.1016/j.pbb.2006.02.017. Epub 2006 Mar 6. PMID 16581115
- [Background] Gonzales D, Rennard SI, Nides M, Oncken C, Azoulay S, Billing CB, Watsky EJ, Gong J, Williams KE, Reeves KR; Varenicline Phase 3 Study Group. Varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs sustained-release bupropion and placebo for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):47-55. doi: 10.1001/jama.296.1.47. PMID 16820546
- [Background] Jorenby DE, Hays JT, Rigotti NA, Azoulay S, Watsky EJ, Williams KE, Billing CB, Gong J, Reeves KR; Varenicline Phase 3 Study Group. Efficacy of varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs placebo or sustained-release bupropion for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):56-63. doi: 10.1001/jama.296.1.56. PMID 16820547
- [Background] Nides M, Oncken C, Gonzales D, Rennard S, Watsky EJ, Anziano R, Reeves KR. Smoking cessation with varenicline, a selective alpha4beta2 nicotinic receptor partial agonist: results from a 7-week, randomized, placebo- and bupropion-controlled trial with 1-year follow-up. Arch Intern Med. 2006 Aug 14-28;166(15):1561-8. doi: 10.1001/archinte.166.15.1561. PMID 16908788
- See also: Tobacco Use Research Center — http://www.tobaccoresearch.umn.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion + Placebo Varenicline: Order 1: Bupropion + Placebo Varenicline \Varenicline + Placebo Bupropion; Order 2: Varenicline + Placebo Bupropion \Bupropion + Placebo Varenicline
  Bupropion SR: Form: tablet, Dosage, Frequency, Duration: Days 1-3, 150 mg, q.d., Days 4-11, 150 mg, b.i.d.
  Varenicline: Form: tablet, Dosage, Frequency, Duration: Days 1-3, .5 mg, q.d., Days 4-7, .5 mg, b.i.d., Days 8-11, 1 mg, b.i.d.
- Varenicline + Placebo Bupropion: Order 1: Bupropion + Varenicline \Varenicline + Placebo Bupropion; Order 2: Varenicline + Placebo Bupropion \Bupropion + Varenicline
  Bupropion SR: Form: tablet, Dosage, Frequency, Duration: Days 1-3, 150 mg, q.d., Days 4-11, 150 mg, b.i.d.
  Varenicline: Form: tablet, Dosage, Frequency, Duration: Days 1-3, .5 mg, q.d., Days 4-7, .5 mg, b.i.d., Days 8-11, 1 mg, b.i.d.
Period: Overall Study
Arm/Group | Bupropion + Placebo Varenicline | Varenicline + Placebo Bupropion
Started | 60 | 61
Completed | 60 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Upropion + Varenicline: Order 1: Bupropion + Varenicline \Varenicline + Placebo Bupropion; Order 2: Varenicline + Placebo Bupropion \Bupropion + Varenicline
  Bupropion SR: Form: tablet, Dosage, Frequency, Duration: Days 1-3, 150 mg, q.d., Days 4-11, 150 mg, b.i.d.
  Varenicline: Form: tablet, Dosage, Frequency, Duration: Days 1-3, .5 mg, q.d., Days 4-7, .5 mg, b.i.d., Days 8-11, 1 mg, b.i.d.
- Total: Total of all reporting groups
Arm/Group | Bupropion + Placebo Varenicline | Upropion + Varenicline | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (11.2) | 40.2 (11.3) | 39.85 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 30 | 31 | 61
Race/Ethnicity, Customized [Number; unit: Count of particpants]
  White | 56 | 52 | 108
Region of Enrollment [Number; unit: participants]
  United States | 60 | 61 | 121

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Withdrawal and Craving
Description: Subjects were analyzed by how they self reported withdrawal or craved cigarettes during treatment Subjects self reported during study visits along with surveys
Time Frame: Change from Base line to 33 weeks
Population: All efforts were made to contact the PI/study team members, but were unsuccessful. No outcome measure study data are available.
Arm/Group | Bupropion + Placebo Varenicline | Varenicline + Placebo Bupropion
Number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Bupropion + Placebo Varenicline vs Varenicline + Placebo Bupropion; Test type: Other — Two tailed testing; p = 0.07, SAS

ADVERSE EVENTS:
Arm/Group | Bupropion + Placebo Varenicline | Varenicline + Placebo Bupropion
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/61
Other Adverse Events (participants affected / at risk) | 0/60 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No